CLINICAL TRIAL: NCT02103400
Title: Physical Training Program in Patients Hospitalized for Community-acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anderson José, Prof., University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAP2014
Record Dates: First submitted 2014-03-22; First posted 2014-04-03 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Walking; Control Groups; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients hospitalized for community-acquired pneumonia
  Interventions: Other: Experimental group
- Control group (Active Comparator): Patients hospitalized for community-acquired pneumonia
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Exercise Training Group
  Other Names: -heating: exercise of free movement of upper and lower limbs; -stretching: stretching various muscle groups; -cardio training walk: 15 minute walk with a high speed; -peripheral muscle strength: exercises using Theraband (R)
  Arms: Experimental group
Other: Control group — Exercise control group
  Other Names: -chest percussion: manual chest percussion; -vibrocompression: manual therapy to the chest; -cough: request for coughing; -breathing exercises: exercises for lung expansion; -Walk: 15 minutes of light walking
  Arms: Control group

SUMMARY:
Hospitalized patients with community-acquired pneumonia (CAP) have reduced functional capacity, peripheral muscle strength and quality of life. Despite the high incidence and severity has not yet been demonstrated whether a physical training program can change these outcomes. Objectives: To evaluate the effects of an exercise training program in patients hospitalized for CAP, to compare this effects with traditional physical therapy and assess whether the inflammatory markers correlate with the functional status of the patient and type of treatment. Methods: A controlled, prospective, randomized clinical trial. Patients hospitalized for CAP, adults, conscious, hemodynamically stable and independent to walk will be studied. In the first day, a medical history, measured dyspnea, incremental shuttle walk test, Glittre test, measurement of peripheral muscle strength, spirometry, and the application of quality of life questionnaire Shor Form 36 will be held. The measurement of inflammatory markers (C-reactive protein and tumor necrosis factor) will also be held. Patients will be randomized into two groups: one will perform a program of physical training (stretching, active resistance exercises and aerobic exercises) and the other group held the traditional physical therapy (bronchial hygiene, breathing exercises and walking) for eight days. On the tenth day the same assessment will be carried out initially described.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pneumonia
* Must be able to walk
* Time less than 48 hours of hospitalization
* Age above 18 years
* Conscious and oriented
* Hemodynamically stable

Exclusion Criteria:

* Patients with other respiratory diseases
* Osteoarticular or cognitive disorders
* Patients who refuse to participate or complete the procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Glittre test | up to 9 months

SECONDARY OUTCOMES:
Shuttle test | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Simone Dal Corso, PhD, Study Director — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Jose A, Dal Corso S. Inpatient rehabilitation improves functional capacity, peripheral muscle strength and quality of life in patients with community-acquired pneumonia: a randomised trial. J Physiother. 2016 Apr;62(2):96-102. doi: 10.1016/j.jphys.2016.02.014. Epub 2016 Mar 17. PMID 26996093